CLINICAL TRIAL: NCT06808113
Title: Study of Circulating and Molecular Markers Functionally Involved in the Processes of Cachexia, Anorexia and Sarcopenia in Patients With Advanced Non-small Cell Lung Cancer (NSCLC).
Brief Title: Circulating and Molecular Markers Involved in the Processes of Cachexia, Anorexia and Sarcopenia in Patients With NSCLC
Acronym: SARCLUNG
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SARCLUNG; 2021.0156 (Other Grant/Funding Number: Fondazione Cassa di Risparmio Bologna)
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; sarcopenia; cachexia; anorexia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sarcopenia; Cachexia; Anorexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim to evaluate whether some substances produced by muscle or adipose tissue may play a role in the course of the disease by interfering with the effectiveness of therapies.

DETAILED DESCRIPTION:
The study is aimed at patients with NSCLC in whom plasma levels of particular biomarkers will be studied before and after treatment with chemotherapy and immunotherapy or immunotherapy alone.

In particular, the plasma levels of GDF15, FGF21, HN, Activin molecules and microRNAs involved in inflammatory processes, called inflammamiR, in particular of microRNA146, 126, 21, 188, 155, will be studied.

Assessments of cellular markers of leukocyte aging will also be performed (determination of telomere length is a widely used measure of biological aging)

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC in advanced stage (IIIB, IV)
* Patients eligible for the treatment with single-agent immunotherapy (Pembrolizumab), or a chemo-immunotherapy combination among the approved ones for I line
* Obtainment of the informations related to medical history and the possibility to have an adequate follow up
* Obtainment of the informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Patients with psychiatric alterations, neurological diseases or other condistions that could not allow adhesion to study protocol and the obtainment of the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC diagnosis in advanced stage, who are eligibble to receive a treatment with single-agent immunotherapy, or a chemo-immunotherapy combination
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Study of serum levels of molecules functionally involved in cachexia/anorexia and sarcopenia, markers of inflammation and markers of aging in patients with NSCLC | The concentration of the respective molecules between the baseline sample and the sample taken after 3 months of treatment will be compared
  To determine the plasma levels of GDF15, FGF21, some microRNAs involved in inflammatory processes called inflammamiR and to perform the measurement of telomere length in leukocytes in plasma samples of patients with NSCLC before and after treatment with chemotherapy and immunotherapy or immunotherapy alone. The association between variables of clinical interest and plasma levels of the aforementioned molecules will be evaluated. In particular, the association between their plasma levels and body composition expressed as a percentage of fat mass and lean mass and overall-survival (OS) and progression-free survival (PFS) will be evaluated.

SECONDARY OUTCOMES:
Flow cytometric analysis of immunosenescence markers in lymphocytes of patients with NSCLC. | The percentage of the different subpopulations between the baseline sample and the sample taken after 3 months of treatment will be compared.
  The leukocyte subpopulations of interest (cell. T naïve, cell. T of the central memory, cell. T of effector memory, cell. Suppressive Myeloids, cell. NK) will be reported as percentages per sample.
  The association between variables of clinical interest and the percentage of different leukocyte subpopulations will be evaluated.
  The association between percentages of white blood cell subpopulations and OS, PFS will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No